CLINICAL TRIAL: NCT06338007
Title: The Relationship of Preoperative Hand Dynamometer Measurement, Pulmonary Function Tests and Modified Frailty Index With Postoperative Outcomes in Patients Undergoing Lung Resection
Brief Title: Relationship Between Hand Dynamometer Measurements, PFT, and mFI With Postoperative Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulay Ulger, Principal Investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2702
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Complication,Postoperative; Lung Cancer
Keywords: Lung Cancer; postoperative complication; modified frailty index; pulmonary function test; hand grip strength measurement
MeSH Terms: conditions — Postoperative Complications; Lung Neoplasms | interventions — Respiratory Function Tests; Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complications (No): Patients who did not experience any postoperative complications within 90 days.
  Interventions: Device: Hand Dynamometer; Diagnostic Test: Pulmonary Function Test; Other: Modified Frailty Index
- Complications (Yes): Patients who experienced any complications within 90 days after surgery.
  Interventions: Device: Hand Dynamometer; Diagnostic Test: Pulmonary Function Test; Other: Modified Frailty Index

INTERVENTIONS:
Device: Hand Dynamometer — Hand grip strength will be measured using a hand dynamometer. Research has demonstrated that hand grip strength is correlated with muscle strength in the upper extremities, as well as overall body and pulmonary muscle strength.
Diagnostic Test: Pulmonary Function Test — Spirometry is a physiological test that measures the ability to inhale and exhale air relative to time. Spirometry is a diagnostic test of several common respiratory disperses such as asthma and chronic obstructive pulmonary disease (COPD). It is also instrumental in monitoring the progression of various respiratory disorders. The main results of spirometry are forced vital capacity (FVC), forced expiratory volume exhaled in the first second (FEV1), and the FEV1/FVC ratio. Pulmonary Function Test analysis values (FEV1, FVC and FEV1 /FVC) will be used.
  Other Names: Spirometry
Other: Modified Frailty Index — The modified frailty index is a valuable preoperative risk assessment tool that can be used to assess the risk of both morbidity and mortality in patients undergoing surgery. It is calculated based on 11 parameters.

SUMMARY:
The study will take place at SBÜ Ankara Atatürk Sanatorium Training and Research Hospital and will include 100 patients over the age of 40 who are scheduled for lung malignancy surgery after 01 April 2024. Informed consent will be obtained from all patients, who will be assigned a number from 1 to 100.

For patients over 40 years of age who are scheduled to undergo lung malignancy resection surgery, demographic data including age, gender, height, weight, body mass index (BMI), diagnosis, comorbidities, and ASA (American Society of Anaesthesiologist) score will be recorded. In addition, hand grip strength measurement, pulmonary function test, and modified frailty index (a scoring system that includes 11 parameters) will be recorded prior to surgery. Intraoperative and postoperative complications will be documented. The duration of the patient's stay in the intensive care unit, chest tube removal, length of hospital stay, and postoperative complications will also be recorded. A follow-up call will be made to the patient by the responsible researcher 90 days after the operation to inquire about any complications that may have developed within that time frame.

The study aims to investigate the relationship between preoperative hand grip strength measurement, pulmonary function test analysis (PFT), and modified frailty index with the duration of intensive care unit stay, chest tube withdrawal time, hospital stay, and postoperative complications in patients undergoing lung resection due to malignancy.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 40 who will undergo lung resection due to malignancy

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients with missing preoperative measurements
* Patients with missing 90-day follow-up data

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During a 3-month period, we calculated that we needed 91 patients to achieve a 95% confidence level with a margin of error of ±5%. This calculation was based on the assumption that 40% of all surgical patients in our clinic had malignant lung resection. We selected a sample size of 100, taking into account possible non-study factors.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Complication | 90 days
  Complication data for patients who underwent lung resection for malignancy during the 90-day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ÜLGER, specialist, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No